CLINICAL TRIAL: NCT07203170
Title: Evaluating the Effectiveness of Leadership Training for Preventing Risk Factors and Promoting Protective Factors Contributing to Psychological Health
Brief Title: Evaluation of the Readiness Supportive Leadership Training - National Guard
Acronym: RESULT-NG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Leslie Hammer, Associate Director of Applied Research, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HT9425-25-1-0668
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Psychological Distress; Anger Problems; Loneliness
Keywords: Military; Psychological health; Problematic anger; Leadership; Resilience; Training intervention
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This clinical trial uses a cluster-randomized Type I Hybrid design at the military unit level, with a wait-list control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leadership Training Intervention (Experimental): Includes leaders, service members, and their spouse/partners where applicable whose units were randomized to receive the RESULT-NG training
  Interventions: Behavioral: Readiness Supportive Leadership Training for the National Guard (RESULT-NG)
- Wait-list Control (No Intervention): The Waitlist Control Arm serves as a delayed start arm. During months 0-15, the waitlist control arm acts as usual practice/no intervention comparator. During months 16-21 (i.e. after final data collection), the waitlist control warm will receive the intervention.

INTERVENTIONS:
Behavioral: Readiness Supportive Leadership Training for the National Guard (RESULT-NG) — RESULT-NG is a multi-level intervention where leaders receive the training intervention, with evaluation of effects at the subordinate, leader and spouse levels.
  RESULT-NG consists of three distinct but related components: 1) a 60-minute, multimedia, interactive digital-learning training session, 2) a two-week behavior tracking exercise that takes less than 2 minutes/day after the digital learning to put what was learned into practice, and 3) a 60-minute facilitated session, either in person or virtual, with trained staff embedded within the National Guard.
  Arms: Leadership Training Intervention

SUMMARY:
The goal of this randomized clinical trial is to evaluate an intervention aimed at increasing the support leaders in the National Guard provide to their subordinates to promote mental health and well-being and reduce risk factors. Survey data will be collected from leaders, service members (SMs) and spouse/partners to evaluate the training effectiveness.

The primary objective of the trial is to demonstrate efficacy in the NG, including effects on leaders, SMs, and spouse/partners on the following outcomes:

H1: Leaders in the intervention group will demonstrate significant improvements in digital learning effects from pre-test to post-test.

H2: The intervention will significantly decrease SM and Leader reports of problematic anger, loneliness, and psychological distress 6-months and then 12-months post-baseline.

H3: Spouses/partners of SMs in the intervention group will report decreases in problematic anger, loneliness, and psychological distress at 6 and 12 months.

Researchers will compare those in the training intervention group to a wait-list control group.

The leadership training builds on a training evaluated in a previous RCT (NCT04152824) adapting from active duty Army to National Guard, including Air NG, and adding an additional facilitated session component. The intervention will include: (1) a 1-hour digital learning utilizing an interactive and self-paced computer-based training, (2) an behavior tracking exercise, and (3) a 1-hour facilitated session, approximately one month later.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age (adults)
* Employed as a member of the Oregon National Guard (ORNG), including Title 5 and 32 civilians, or is a spouse/partner of an ORNG service member married or cohabitating with the SM for 6 months or more

Exclusion Criteria:

* Under 18 years of age
* Not employed as a member of the Oregon National Guard (ORNG), including Title 5 and 32 civilians, or is a spouse/partner of an ORNG service member married or cohabitating with the SM for less than 6 months

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5400 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Dimensions of Anger (DAR-5) | 0 months, 6 months, and 12 months
  Each item in the scale uses a 5-point Likert scale (1 = none of the time, 2 = a little of the time, 3 = some of the time, 4 = most of the time, and 5 = all of the time). A cutoff score of 8 or greater on the DAR-3 is considered indicative of problematic anger and shows optimal sensitivity and specificity.
Depression Subscale- Primary Health Questionnaire (PHQ-9) | 0 months, 6 months, and 12 months
  Nine item questionnaire based on the diagnostic criteria for major depressive disorder in the DSM-5. Each question is scored on a scale of 0 to 3, with higher scores indicating greater symptom severity.
Brief Loneliness Scale | 0 months, 6 months, and 12 months.
  3-item scale. Responses are summed to calculate a total score between 3 and 9. Lower scores (3-5) indicate less loneliness, while higher scores (6-9) suggest more significant feelings of loneliness.

IPD SHARING:
Plan to Share IPD: Yes
All deidentified IPD collected throughout the trial.
Supporting Information: Study Protocol
URL: https://nda.nih.gov/